CLINICAL TRIAL: NCT03589287
Title: A Phase I/IIa Clinical Study of Treatment for Knee Osteoarthritis by Intra-articular Injection of Allogeneic Bone Marrow Derived Mesenchymal Stem Cells.
Brief Title: Allogeneic Bone Marrow MSC Therapy for Knee Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Virginia Contract Research Organization Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2016-11-006C
Record Dates: First submitted 2018-06-04; First posted 2018-07-17 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Knee Osteoarthritis
Keywords: Intra-articular (IA), Allogeneic, MSC, OA
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The treatment protocol consists of two stages: the first stage is a traditional 3+3 dose-escalation open study design with three cohorts. At the second stage, a total of 6 patients with knee OA will be treated by the cell products of the maximum tolerance dose (MTD) as determined by the results of the first stage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chondrochymal® 1 x 10^7 cells (Experimental): At this stage, 3 patients with knee OA will be treated by the cell products of this dose.
  Interventions: Biological: Chondrochymal®
- Chondrochymal® 5 x 10^7 cells (Experimental): At this stage, 3 patients with knee OA will be treated by the cell products of this dose.
  Interventions: Biological: Chondrochymal®
- Chondrochymal® 10 x 10^7 cells (Experimental): At this stage, 3 patients with knee OA will be treated by the cell products of this dose.
  Interventions: Biological: Chondrochymal®

INTERVENTIONS:
Biological: Chondrochymal® — Allogeneic Bone Marrow Derived Mesenchymal Stem Cells

SUMMARY:
The Clinical trial is a phase I/IIa clinical study for treatment of knee osteoarthritis by intra-articular injection of bone marrow derived allogeneic mesenchymal stem cells. Primary endpoint of the study is safety of allogeneic BM-MSCs application on knee OA with single dose IA injection and the MTD. Secondary endpoint is the effect of allogeneic BM-MSCs transplantation including clinical and image observation since the MSCs have multi-lineage differentiation potential such as chondrocyte differentiation, anti-inflammation and immune-modulation.

DETAILED DESCRIPTION:
Osteoarthritis of the knee (Knee Osteoarthritis, Knee OA) is a joint disease that primarily affects cartilage. Cartilage is the smooth tissue covering the ends of bones within the joint. In people who suffer from knee OA, articular cartilage top is broken down and worn away, resulting in the underlying bones to rub against each other. This friction can cause pain, joint swelling and decreased range of motion (ROM). Eventually, the joint may become deformed and bone spurs may form around the edges. With the advances in biotechnology, cell therapy in the application of cartilage reconstruction has gradually matured. The purpose of this study is to assess the safety and efficacy of single intra-articular (IA) injection of allogeneic bone marrow (BM) mesenchymal stem cells (MSCs) for knee OA. The same cell products used in this trial have been applied in a phase I/IIa clinical trial in Taiwan for the treatment of critical limb ischemia, and so far no treatment-related adverse effect has been observed. In the current trial, allogeneic bone marrow MSCs of up to 4 donors will be isolated. BM MSCs are expanded and applied for a phase I/IIa study in treating 15-24 recipient patients with knee OA. The treatment protocol consists of two stages: the first stage is a traditional 3+3 open dose-escalated study design with three cohorts of dosing groups: (1) 1 x 10^7 cells, (2) 5 x 10^7 cells and (3) 10 x 10^7 cells. At the second stage, knee OA patients will be treated by the cell products of the maximum tolerance dose (MTD) as determined by the results of the first stage. All the study subjects will be followed up to 6 months (24 weeks) after the treatment for safety and preliminary efficacy evaluation, which the latter will include both clinical and imaging study assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 40 years old, completing the informed consent process for participating the clinical trial
2. Patients diagnosed with unilateral/bilateral knee osteoarthritis of grade II, III and IV (Kellgren and Lawrence scale) as assessed by doctors, who are not suitable for, or not willing to undergo knee surgery (including total knee replacement)
3. Pain of the knee as assessed by visual analogue scale (VAS) to be 4 or higher (VAS ≥ 4)
4. Body mass index (BMI) between 20 and 35 kg/m2
5. Neither local/systemic bacteremia nor acute infection around the knee joint

Exclusion Criteria:

1. Physiologically or psychologically inappropriate for participating the trial as evaluated by the investigators
2. Patients with congenital or acquired bone hypoplasia (Varus more than 10o or Valgus more than 20o)
3. BMI less than 20 or more than 35 (Class II obesity)
4. Female who is pregnant or breastfeeding, or in childbearing age; male or female subjects who are not able to use appropriate contraception methods during the trial
5. Patients with muscular or neurological diseases causing deformity of the targeted knee joint(s), which might interfere with the evaluation of trial.
6. Patients with malignant tumors, or benign tumors that may interfere with the trial treatment or subsequent evaluation.
7. Immunocompromised or patients suffering from immune diseases under long-term immuno-suppressive medication such as steroids, however, topical steroid is not included
8. Patients with coagulation or hematological disorders not suitable for intra-articular (IA) injection
9. Known or possible allergy to components in the product under trial
10. Patients had any IA injection or surgery of the targeted knee within the last 3 months
11. Patients with crippled lower limbs rated ACR functional class IV (Largely or Wholly Incapacitated) or cannot walk without one/two arms-operated walking assisting device (defined by CNS15390)
12. Spontaneous knee osteonecrosis
13. Previous surgery of the knee that may cause metal imaging artifacts on imaging study
14. Patients have claustrophobia and/or cannot take magnetic resonance imaging (MRI) test
15. Any metal devices placed in the body such as pacemaker, artificial heart valve, or hemostatic clamps/clips for intracranial aneurysm posing risk under magnetic field (of MRI)
16. Patients with severe unilateral (or bilateral) knee osteoarthritis who have decided to receive surgery (including total knee replacement) on the affected knee (or both knees if bilateral) after advised by their surgeon.
17. Having participated other clinical trials with medications (including cellular therapy) within the past 3 months prior to subject screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as measure of safety and tolerability | 24 weeks
  treatment-related adverse events assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Efficacy - Radiographic evidence | 24 weeks
  Change in cartilage thickness of the knee using MRI and X-ray
Efficacy - WOMAC assessment | 24 weeks
  Change in joint function from baseline WOMAC assessment
Efficacy - Visual Analogue Scale(VAS) assessment | 24 weeks
  The Visual Analog Scale (VAS) is a unidimensional measure of pain intensity. The scale is most commonly anchored by "no pain " (score of 0) and "worst imaginable pain" (score of 10).
Efficacy - Lequesne Index assessment | 24 weeks
  Change in arthritis pain scores on the Lequesne Index
Efficacy - Keen Society Score(KSS) assessment | 24 weeks
  The knee society score is divided into four parts: it consists of the ''Symptoms''(25 points), the ''Patient satisfaction''(40 points), the ''Patient expectation''(15 points) and the ''Functional activities''(100 points). Each part will be evaluated separately.
Efficacy - QOL assessment | 24 weeks
  Change in scores on the QOL

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chau Chang, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan